CLINICAL TRIAL: NCT04143022
Title: Evaluation of the Effects of Acupuncture Press Needle in Mild to Moderate Obstructive Sleep Apnea Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201801807A3
Record Dates: First submitted 2019-03-20; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-01

CONDITIONS: Apnea, Obstructive Sleep; Snoring
Keywords: acupuncture press needle; obstructive sleep apnea; polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Intervention Model Description: 40 eligible participants diagnosed as mild to moderate OSA will be enrolled and randomly allocated to group A and group B. Press needle will be applied to acupoints at Jin's 3-tongue point ( EX-HN21 and the two extra channel points, 0.8 individual cun lateral to both sides of EX-HN21) and EX-HN25 in group A and at EX-CA1, EX-CA5 and EX-CA6 in group B. Each subject will start first course and receive the treatment 2 times a week for 4 weeks (8 times in total). Then, it takes 2-week washout period and make group A and group B crossover. Second course begins after 2-week washout period with the same treatment times as the first course. The primary outcomes include the apnea-hypopnea index (AHI), snore time, snore index assessed by polysomnography, snore sound assessed by SnoreLab (snore recording and analysis application), and secondary outcome includes snore outcome survey questionnaire (SOS).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (acupuncture press needle) (Active Comparator): Group A subjects first receive acupuncture press needle treatment at acupoint of Jin's 3-tongue point and EX-HN25. Then, it takes 2-week washout period. After washout period, subjects receive another course of treatment at acupoint of EX-CA1, EX-CA5 and EX-CA6. Each subject receive 2 times a week of treatment for 4 weeks (8 times in total) in each course.
  Interventions: Device: acupuncture press needle
- group B (acupuncture press needle) (Active Comparator): Group B subjects first receive acupuncture press needle treatment at acupoint of EX-CA1, EX-CA5 and EX-CA6. Then, it takes 2-week washout period. After washout period, subjects receive another course of treatment at acupoint of Jin's 3-tongue point and EX-HN25. Each subject receive 2 times a week of treatment for 4 weeks (8 times in total) in each course.
  Interventions: Device: acupuncture press needle

INTERVENTIONS:
Device: acupuncture press needle — Press needle will be applied to acupoints at Jin's 3-tongue point ( EX-HN21 and the two extra channel points, 0.8 individual cun lateral to both sides of EX-HN21) and EX-HN25 in group A and at EX-CA1, EX-CA5 and EX-CA6 in group B. Each subject will start first course and receive the treatment 2 times a week for 4 weeks (8 times in total). Then, it takes 2-week washout period and make group A and group B crossover. Second course begins after 2-week washout period with the same treatment times as the first course.

SUMMARY:
The aim of this study is to investigate the effects of acupuncture press needle in mild to moderate obstructive sleep apnea patients.

DETAILED DESCRIPTION:
Obstructive sleep apnea(OSA) is characterized by multiple episodes of upper airway collapse during sleep and considered as a major health issue worldwide due to comorbidity with obesity, hypertension, diabetes and more advanced cardiovascular diseases. The noisy sounds of snoring caused by OSA bother bed partner sleepless and lead to long-term health problems. Most patients do not tolerate nasal continuous positive airway pressure device, which is the gold standard treatment of OSA. Press needle is one kind of acupuncture which possesses more safety and convenient, few complications and prolonged period of treatment time compared to conventional acupuncture. To date, there is no study to evaluate the effects of press needle in treating OSA. The investigators hypothesize that press needle is effective with high acceptability among OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign inform consent with aged more than 20 years old
* Mild to moderate OSA, AHI < 30

Exclusion Criteria:

* Severe OSA, AHI > 30
* Significant lung disease
* Skeletal facial framework problems
* Central apnea
* Undergone oropharyngeal operations, continuous positive airway pressure or oral devices
* Taking hypnotic drugs
* Pregnancy or breast-feeding
* Receiving acupuncture in recent 2 weeks

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-23 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-22 (Estimated)

PRIMARY OUTCOMES:
Change of Apnea-Hypopnea Index (AHI) measured by polysomnography (PSG) | change from baseline AHI at 4 weeks and 10 weeks post-treatment
  PSG is a multi-parametric test used in the study of sleep and as a diagnostic tool in sleep medicine. AHI is calculated by dividing the number of apnea events by the number of hours of sleep.
Change of Snore Index (SI) measured by polysomnography (PSG) | change from baseline SI at 4 weeks and 10 weeks post-treatment
  PSG is a multi-parametric test used in the study of sleep and as a diagnostic tool in sleep medicine. SI is calculated by dividing the number of snore events by the number of hours of sleep.

SECONDARY OUTCOMES:
Change of snore outcome survey questionnaire (SOS) | change from baseline Snore outcome survey questionnaire (SOS) at 4 weeks and 10 weeks post-treatment
  The questionnaire used for a patient-based measure for the full range of sleep-disordered breathing patients in whom snoring is a primary symptom, where the goal is to measure the snoring component of sleep-disordered breathing. Total scores are normalized on a scale from 0 to 100. Higher values indicates a better outcome.
Change of anti-snore solution record (apnea counts and snore counts) | This application is applied for every night to record apnea counts and snore counts before treatment and last for 10 weeks.
  Anti-snore solution is one kind of smartphone application for recording sleep condition. Apnea counts and sleep counts can be detected by this software.
Change of anti-snore solution record (snore volume) | This application is applied for every night to record snore volume before treatment and last for 10 weeks.
  Anti-snore solution is one kind of smartphone application for recording sleep condition. Snore volume (in dB) can be detected by this software.

CONTACTS AND LOCATIONS:
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No
1. There will be a research number representing the identity. This number will not display the name, identification number, and address.
  2. For the results and diagnosis of the visit, the research host will maintain a confidential attitude and carefully maintain the privacy. If research results are published, the identity will remain confidential.
  3. Please also understand that if the participant signs the consent form, the participant agrees that the visit record can be directly reviewed by the monitor, auditor, research ethics committee and the competent authority to ensure that the research process and data comply with relevant laws and regulations. These people also promise not to violate the confidentiality of your identity.